CLINICAL TRIAL: NCT02009150
Title: Evaluation of REAL IMAGING'S 3D Functional Metabolic Imaging and Risk Assessment ("3D MIRA") System in Women at High Risk for Breast Cancer
Brief Title: Evaluation of a Novel Infra-red Breast Imaging System for Risk Assessment in Women at High Risk for Breast Cancer.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Real Imaging Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 960-CSP-ISR_HighRiskMC_ILS1
Record Dates: First submitted 2013-12-07; First posted 2013-12-11 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Women at high risk for breast cancer: Proven carriers of deleterious BRCA1 or BRCA2 mutations Or Women that were found to have a lifetime risk of developing breast cancer greater or equal to 20% based on Tyrer-Cuzick, Gail or Clause risk models.

SUMMARY:
Three-dimensional functional Metabolic Imaging (3D MIRA) is a new infrared imaging technology using the Real Imager 4(RI4) developed by Real Imaging. This technology generates 3D metabolic maps and based on sophisticated machine learning technology, provides objective risk assessment for the presence of malignant tumor. The procedure is non-invasive, comfortable and does not involve ionizing radiation. Moreover, Real Imaging's 3D Functional MIRA is unaffected by breast density and is therefore ideal for evaluating patients with mammographically dense breasts.

The purpose of this clinical study is to assess the ability of this novel technology to detect clinically occult breast cancer in a cohort of women that are at high risk for breast cancer.

We hypothesize that the combination of screening mammography and metabolic screening (3D MIRA) will result in significantly higher breast cancer detection rates.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Woman has read, understood and signed the inform consent form
* Age: 20 years and older
* Women who are asymptomatic for breast cancer
* Proven carriers of deleterious BRCA1 or BRCA2 mutations Or Women that were found to have a lifetime risk of developing breast cancer greater or equal to 20% based on Tyrer-Cuzick, Gail or Clause risk models
* Women scheduled to undergo routine mammography and/or US or MRI screening

Exclusion Criteria:

* Women who have had a mammography and/or ultrasound examination performed on the day of the study prior to MIRA scan
* Women who had a lumpectomy surgery
* Women who had undergone mastectomy and/or reconstruction
* Women who have undergone any type of breast surgery throughout the 6 months preceding the study
* Women who have had a breast biopsy performed throughout the 10 weeks preceding the study.
* Women who have a fever on the day of the MIRA imaging
* Women who are pregnant
* Women who are breast-feeding
* Women who had undergone breast reduction/augmentation

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who are determined to have high risk of breast cancer and who are screened biannually by existing screening modalities (mammography, ultrasound or MRI)
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of 3D MIRA as a breast imaging aid in women with a high risk of breast cancer | up to 36 months

SECONDARY OUTCOMES:
To test whether repetitive screening with 3D MIRA technology can provide information on the likelihood of developing breast cancer. | up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Miri Sklair-Levy, MD, Principal Investigator — The Chaim Sheba Medical center at Tel-Hashomer
Locations (1):
- The Chaim Sheba Medical Center at Tel-Hashomer, Ramat Gan, Israel